CLINICAL TRIAL: NCT03644095
Title: A Phase I, Open-label, Single-dose, Randomized, 2-way Crossover Bioequivalence Study Comparing Mucinex® SE Extended-Release 600 mg Bi-layer Tablet to a Reference Immediate-Release Guaifenesin 600 mg (Taken as 200 mg q4h) in Normal Healthy Subjects.
Brief Title: Bioequivalence Study Comparing Mucinex Extended-release 600 mg Tablets to Immediate-release Guaifenesin 600 mg in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Inc. (Industry)
Responsible Party: Sponsor
Organization: Reckitt Benckiser LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-GGE-02
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Guaifenesin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mucinex® SE 600 mg (extended-release) (Experimental): Single dose of Mucinex® SE extended-release 600 mg bi-layer tablet taken with 240 mL of water after an overnight fast
  Interventions: Drug: Mucinex® SE
- Vicks Cough Syrup 200 mg (Active Comparator): Vicks Cough Syrup for Chesty Coughs 200 mg every 4 hours taken with 240 mL of water after an overnight fast
  Interventions: Drug: Vicks Cough Syrup for Chesty Coughs

INTERVENTIONS:
Drug: Mucinex® SE — Single dose of Mucinex® SE extended-release 600 mg bi-layer tablet
  Other Names: guaifenesin bi-layer tablet
  Arms: Mucinex® SE 600 mg (extended-release)
Drug: Vicks Cough Syrup for Chesty Coughs — Vicks Cough Syrup for Chesty Coughs 15 mL (200 mg guaifenesin q4h) immediate release (IR) syrup
  Other Names: guaifenesin
  Arms: Vicks Cough Syrup 200 mg

SUMMARY:
Determine bioequivalence, safety and tolerability of guaifenesin extended-release 600 mg (Mucinex® SE) compared to an immediate-release syrup reference product in normal healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females between the ages of 19 and 55 years, inclusive.
2. Females of childbearing potential must be using one of the following acceptable birth control methods:

   1. Intra-uterine device in place for at least 3 months prior to Day 1 of Period 1 through 30 days beyond study completion;
   2. Barrier method (condom or diaphragm) with spermicide for at least 7 days prior to screening through 30 days beyond study completion;
   3. Stable hormonal contraceptive (e.g., oral, depo injection, transdermal patch, or vaginal ring) for at least 3 months prior to Day 1 of Period 1 through 30 days beyond completion of study;

   Abstinence is not an acceptable form of contraception; however, abstinent female subjects may be admitted to the study if they agree, and have signed a statement to the effect, that upon becoming sexually active, will use a condom with spermicide from screening through 30 days beyond completion of the study.
3. Females of non-childbearing potential should be surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to study or hysterectomy and/or bilateral oophorectomy at least 3 months prior to Day 1 of Period 1) or postmenopausal >2 years prior to Day 1 of Period 1. A follicle stimulating hormone (FSH) concentration >40 miU/mL must be obtained and recorded for any postmenopausal females.
4. Good general health as determined by the Principal Investigator's (PI) review of medical history, physical examination, vital sign measurements, electrocardiogram (ECG), and clinical laboratory measures.
5. Body weight between 50 - 100 kg and body mass index (BMI) within 18 - 30 kg/m2.
6. Non-tobacco users, who have not used nicotine or nicotine-containing products for at least 365 days prior to Day 1 of Period 1.
7. Able to read, understand and sign the informed consent after the nature of the study has been explained.
8. Negative urine screen for drugs of abuse and alcohol at screening and each check in.
9. If female, negative finding on serum pregnancy test at screening and each check-in.
10. Non alcohol or drug abuser - non alcohol abuse is defined as history of less than 4 drinks daily. A drink is defined as 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of spirits (i.e., 'hard' liquor such as gin, whiskey, or vodka).

Exclusion Criteria:

1. Clinically significant abnormalities detected by medical history, physical examination, vial sign measurements, ECG, or clinical laboratory findings (as determined by the PI/designee) including a hemoglobin value <12 gm/dL at screening. If a subject's hemoglobin drops below 11.0 gm/dL during the study, the subject may be dropped from the study at the discretion of the PI.
2. Any disease or condition, which could impact absorption, distribution, metabolism, or elimination of the study drugs (as determined by the PI/designee).
3. Females who are pregnant or nursing.
4. History of sensitivity reaction to guaifenesin.
5. Receipt of an investigational drug within 30 days prior to Day 1 of Period 1.
6. Abnormal diet (for whatever reason) during the 30 days prior to Day 1 of Period 1.
7. Donation of blood or significant loss of blood within 56 days or plasma within 14 days prior to Day 1 of Period 1.
8. Known or suspected use of illicit drugs.
9. The use of any medication (with the exception of hormonal contraceptives for women of childbearing potential) for 14 days or 5 half-lives of the drug (whichever is longer) prior to Day 1 of Period 1.
10. Test positive for Hepatitis B surface antigen, Hepatitis C antibodies, or HIV at Screening.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01-16 (Actual); Primary Completion 2009-02-01 (Actual); Study Completion 2009-02-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-centre study.
Pre-assignment Details: Total 30 subjects were enrolled in the study and all 30 subjects completed the study.
Groups:
- Mucinex First, Then Vicks: Treatment Sequences 1: Treatment A in Period 1, then Treatment B in Period 2
  Test (Treatment A): Subjects received a single PO dose of 1 Mucinex® 600 mg guaifenesin ER bi-layer tablet administered with 240 mL of water.
  Reference (Treatment B): Subjects received a single PO dose of 15 mL (200 mg) Vicks Cough Syrup for Chesty Coughs Containing Guaifenesin every 4 hours (q4h) x 3 doses each administered with 240 mL of water.
  There was a 7 days washout period between each administration.
- Vicks First, Then Mucinex: Treatment Sequences 2: Treatment B in Period 1, then Treatment A in Period 2
  Reference (Treatment B): Subjects received a single PO dose of 15 mL (200 mg) Vicks Cough Syrup for Chesty Coughs Containing Guaifenesin every 4 hours (q4h) x 3 doses each administered with 240 mL of water.
  Test (Treatment A): Subjects received a single PO dose of 1 Mucinex® 600 mg guaifenesin ER bi-layer tablet administered with 240 mL of water.
  There was a 7 days washout period between each administration.
Period: Period 1
Arm/Group | Mucinex First, Then Vicks | Vicks First, Then Mucinex
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | Mucinex First, Then Vicks | Vicks First, Then Mucinex
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Mucinex First, Then Vicks | Vicks First, Then Mucinex
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Test (Treatment A): Subjects received a single PO (by mouth) dose of 1 Mucinex® 600 mg guaifenesin ER bi-layer tablet administered with 240 mL of water.
  Reference (Treatment B): Subjects received a single PO (by mouth) dose of 15 mL (200 mg) Vicks Cough Syrup for Chesty Coughs Containing Guaifenesin every 4 hours (q4h) x 3 doses each administered with 240 mL of water.
  Period 1: Treatment A or Treatment B at Sequence AB
  Period 2: Treatment B or Treatment A at Sequence BA
  There was a 7 days washout period between each administration.
Arm/Group | Overall Study
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.5 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27
  Hispanic | 3
Weight [Mean (Standard Deviation); unit: lb] | 162.2 (25.37)
Height [Mean (Standard Deviation); unit: In] | 68.92 (4.062)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 23.937 (2.6486)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Guaifenesin
Description: Pharmacokinetic Parameter (Cmax) Maximum observed plasma concentration.
Time Frame: 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14, 16 and 24 hours (post-dose) on Day 1 and 2
Population: The Pharmacokinetic (PK) parameters were calculated from individual plasma concentration-time data (using actual blood draw times).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Test (Treatment A): Test (Treatment A): Subjects received a single PO dose of 1 Mucinex® 600 mg guaifenesin ER bi-layer tablet administered with 240 mL of water.
- Reference (Treatment B): Reference (Treatment B): Subjects received a single PO dose of 15 mL (200 mg) Vicks Cough Syrup for Chesty Coughs Containing Guaifenesin every 4 hours (q4h) x 3 doses each administered with 240 mL of water.
Arm/Group | Test (Treatment A) | Reference (Treatment B)
Number analyzed (Participants) | 30 | 30
ng/mL | 857 (469) | 1390 (575)

2. Primary Outcome: Area Under Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUC(0-t)) of Guaifenesin
Description: Area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration, as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Population: PK Data Set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Test (Treatment A) | Reference (Treatment B)
Number analyzed (Participants) | 30 | 30
ng*hr/mL | 3404.7 (1661.1) | 4447.1 (1627.4)

3. Primary Outcome: Area Under Plasma Concentration-time Curve From Time 0 to Infinity (AUC(0-inf)) of Guaifenesin
Description: Area under the plasma concentration versus time curve from time 0 to infinity, calculated as AUC 0-t + C last/kel, where C last is the last measurable concentration and kel is the apparent first-order terminal elimination rate constant.
Time Frame: as for outcome 1
Population: PK Data Set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Test (Treatment A) | Reference (Treatment B)
Number analyzed (Participants) | 30 | 30
ng*hr/mL | 3442.0 (1674.8) | 4456.4 (1630.7)

4. Primary Outcome: Time to Maximum Observed Concentration (Tmax) of Guaifenesin
Description: Pharmacokinetic Parameter (Tmax) Time of the maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: PK Data Set
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Test (Treatment A) | Reference (Treatment B)
Number analyzed (Participants) | 30 | 30
hr | 0.885 (0.537) | 3.05 (2.47)

5. Primary Outcome: Area Under Plasma Concentration Curve Ratio (AUCR) of Guaifenesin
Description: Pharmacokinetic Parameter AUCR is the ratio of AUC(0-t) to AUC(0-inf). AUCR = AUC(0-t) / AUC(0-inf)
Time Frame: as for outcome 1
Population: PK Data Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Test (Treatment A) | Reference (Treatment B)
Number analyzed (Participants) | 30 | 30
Ratio | 0.988 (0.0144) | 0.998 (0.00167)

6. Primary Outcome: Apparent Terminal Elimination Rate Constant (Kel) of Guaifenesin
Description: Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma concentration versus time curve. The parameter was calculated by linear least-squares (LS) regression analysis using the maximum number of points (e.g. 3 or more non-zero plasma concentrations) in the terminal log-linear phase.
Time Frame: as for outcome 1
Population: PK Data Sets
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Test (Treatment A) | Reference (Treatment B)
Number analyzed (Participants) | 30 | 30
1/hr | 0.373 (0.181) | 0.716 (0.110)

7. Primary Outcome: Apparent Terminal Elimination Half-life (t1/2) of Guaifenesin
Description: Apparent first-order terminal elimination half-life, calculated as ln(2)/kel.
Time Frame: as for outcome 1
Population: PK Data Set
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Test (Treatment A) | Reference (Treatment B)
Number analyzed (Participants) | 30 | 30
hr | 2.26 (0.948) | 0.989 (0.147)

8. Secondary Outcome: Number of Adverse Events (AE) of Participants
Description: Mild = AE does not limit usual activities;subject may experience slight discomfort; Moderate = AE results in some limitation of usual activities; subject may experience significant discomfort; Severe = AE results in an inability to carry out usual activities; Probable = Most likely that the AE was caused by study drug; Possible = Reasonable suspicion that the AE was caused by the study drug; Unlikely = Slight but remote chance that the AE was caused by study drug but the balance of judgment is that it was most likely not due to the study drug.
Time Frame: Upto Day 2
Measure: Number; unit: Events
Arm/Group | Test (Treatment A) | Reference (Treatment B)
Number analyzed (Participants) | 30 | 30
Events
  TEAE by severity: Mild | 7 | 8
  TEAE by severity: Moderate | 0 | 0
  TEAE by severity: Severe | 0 | 0
  Relationship to Drug: Probable | 0 | 0
  Relationship to Drug: Possible | 6 | 3
  Relationship to Drug: Unlikely | 1 | 5

ADVERSE EVENTS:
Time Frame: Up to Day 17
Arm/Group | Test (Treatment A) | Reference (Treatment B)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 6/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (Treatment A) (N=30) | Reference (Treatment B) (N=30)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No